CLINICAL TRIAL: NCT05674344
Title: Calibration and Validation of the Masimo Rad-G With Temperature Device in Febrile Patients
Brief Title: Calibration and Validation of the Masimo Temperature Device in Febrile Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHOC0008
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Masimo noninvasive temperature device (Experimental): All subjects who qualify for the trial and participate in data collection will have temperature taken using the Masimo noninvasive temperature device and the reference temperature device.
  Interventions: Device: Masimo Temperature device

INTERVENTIONS:
Device: Masimo Temperature device — Non-invasive temperature device

SUMMARY:
The goal of this clinical trial is to test the performance of the Masimo noninvasive temperature device in patients with fever. The main question it aims to answer is whether the Masimo temperature device is comparable to standard methods of taking temperature such as inserting a probe under the tongue or using a forehead thermometer.

Participants will be asked to sit still while rounds of measurements are taken using the Masimo temperature device and the reference temperature device. Researchers will compare the measurements taken with the Masimo device with the measurements taken with the reference device.

DETAILED DESCRIPTION:
Individual sites are only representative of a subset of the overall population, per ISO 80601-2-56:2017(Medical electrical equipment - Part 2-56: Particular requirements for basic safety and essential performance of clinical thermometers for body temperature measurement), and therefore clinical bias and limits of agreement should not be evaluated for the subsets. Publication of results should include repeatability from individual sites and the combined clinical bias and limits of agreement (NCT05787782, NCT05674344, and NCT05779397)

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 1year old
* Febrile at time of enrollment: ≥ 99.5oF/37.5oC for patients ages 1-5 years; ≥ 100.4oF/38oC for patients older than 5 years old.
* English- or Spanish-speaking patient or parent/LAR

Exclusion Criteria:

* Patients deemed not suitable for the study at the discretion of the investigator
* Patients who are rated as a 1 or 2 Emergency Severity Index

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 1, Orange, California, United States

REFERENCES:
- See also: NCT05787782, Validation of the Masimo INVSENSOR00063 in Febrile and Afebrile Subejcts — https://clinicaltrials.gov/ct2/show/NCT05787782?term=koei0004&draw=2&rank=1
- See also: NCT05779397, Clinical Performance of Masimo Rad-GT — http://clinicaltrials.gov/ct2/show/NCT05779397?term=CIP-1064&draw=2&rank=1

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Masimo Noninvasive Temperature Device
Started | 170
Completed | 146
Not Completed | 24
Not completed — Screen Fail | 21
Not completed — Incomplete study procedures | 3

BASELINE CHARACTERISTICS:
Arm/Group | Masimo Noninvasive Temperature Device
Number analyzed (Participants) | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 170
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 126
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 92
  More than one race | 0
  Unknown or Not Reported | 65
Region of Enrollment [Number; unit: participants]
  United States | 170

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Masimo RAD-GT Temperature Measurments
Description: The accuracy of the Masimo Rad-GT sensor will be determined by calculating the clinical bias (Δcb), limits of agreement (LA), and repeatability (σr). The temperature measurements from Masimo Rad-GT will be compared to the reference temperature measurements (degrees Celsius).
Time Frame: 15-30 Minutes
Population: Subject 1 to 91 were part of the calibration phase of the study (91 subjects) and data was excluded from analysis.
  14 excluded due to screen fails.
  Subject 92 to 170 (79 subjects) were part of the validation phase of the study. 10 screen fails. 4: Any subject who does not complete at least one full round of measurements. 26: Any subject whose data suggests existence of external conditions that interfere with RCT (reference clinical thermometer) or Rad-GT measurements.
Measure: Number; unit: Degrees Celsius
Arm/Group | Masimo Noninvasive Temperature Device
Number analyzed (Participants) | 39
Degrees Celsius
  Clinical Bias | -0.24
  Limits of Agreement | 0.85
  Repeatability | 0.09

ADVERSE EVENTS:
Time Frame: Approximately 15-30 minutes during data collection
Arm/Group | Masimo Noninvasive Temperature Device
All-Cause Mortality (participants affected / at risk) | 0/170
Serious Adverse Events (participants affected / at risk) | 0/170
Other Adverse Events (participants affected / at risk) | 0/170

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT05674344/Prot_SAP_000.pdf